CLINICAL TRIAL: NCT01957644
Title: An Open Label Phase I Dose Escalation Trial to Investigate the Maximum Tolerated Dose, Safety, Pharmacokinetics and Efficacy of Intravenous Volasertib in Combination With Subcutaneous Azacitidine in Patients With Previously Untreated High-risk Myelodysplastic Syndrome (MDS) or Chronic Myelomonocytic Leukemia (CMML) and Not Candidates for Haematopoetic Stem Cell Transplant
Brief Title: Phase I Dose Escalation Trial of Volasertib in Combination With Azacitidine in Patients With MDS or CMML
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1230.33; 2013-001290-24 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-10-01; First posted 2013-10-08 (Estimated); Results first posted 2019-02-08 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2018-09

CONDITIONS: Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — Azacitidine; BI 6727

ARMS (3):
- Schedule A (Experimental): Volasertib (d1 - one hour iv.) + Azacitidine 75 mg/m2 once daily on Days 1-7 (7 consecutive days) (28-day cycle)
  Interventions: Drug: Azacitidine; Drug: Volasertib
- Schedule B (Experimental): Volasertib (d 7 - one hour iv.) + Azacitidine 75 mg/m2 once daily on Days 1-7 (7 consecutive days) (28-day cycle)
  Interventions: Drug: Azacitidine; Drug: Volasertib
- Schedule C (Experimental): Volasertib (d 1 and 7 - one hour iv.) + Azacitidine 75 mg/m2 once daily on Days 1-7 (7 consecutive days) (28-day cycle)
  Interventions: Drug: Azacitidine; Drug: Volasertib

INTERVENTIONS:
Drug: Azacitidine
Drug: Volasertib

SUMMARY:
To investigate the maximum tolerated dose (MTD), safety, pharmacokinetics, and efficacy of volasertib in combination with azacitidine in patients with myelodysplastic syndromes (MDS) or chronic myelomonocytic leukemia (CMML) and not candidates for hematopoietic stem cell transplant

ELIGIBILITY:
Inclusion criteria:

* Adult patients with previously untreated, intermediate-2 or high- risk MDS or CMML not eligible for hematopoietic stem cell transplantation (HSCT) based on documented patients characteristics like age, performance status, concomitant diagnoses, and organ dysfunctions
* Further inclusion criteria apply

Exclusion criteria:

* Prior or concomitant therapy for higher risk MDS (for example, but not limited to, hypomethylating agents like azacitidine). Note: Prior treatment with erythropoetin (EPO) is allowed up to > 1 week before treatment with study medication. Patients must have not received MDS therapy since diagnosis of higher-risk MDS. However, previous lenalidomide treatment could have been administered for lower-risk MDS treatment as long as this therapy was discontinued at least > 4 weeks before initiation of the current study treatment.
* Treatment with any investigational drug within 2 weeks before first administration of present trial drug or within less than 5 half lives of the investigational drug before treatment with the present trial drug, whichever is longer.
* Second malignancy currently requiring active therapy (except for hormonal/anti-hormonal treatment, e.g. in prostate or breast cancer).
* Corrected QT interval according to Fridericia (QTcF) prolongation > 470 ms or QT prolongation deemed clinically relevant by the investigator (e.g., congenital long QT syndrome).The QTcF will be calculated as the mean of the 3 Electrocardiograms (ECGs) taken at screening.
* Total bilirubin > 1.5 x upper limit of normal not related to Gilberts disease, hemolysis, or secondary to MDS.
* Aspartate amino transferase (AST) or alanine amino transferase (ALT) > 2.5 x the upper limit of normal (ULN) Creatinine > 1.5 x ULN
* Active hepatitis B or hepatitis C, or laboratory evidence for a chronic infection (hepatitis test results done in routine diagnostics are acceptable if done within 14 days before first study treatment dose).
* HIV infection (HIV test results in routine diagnostics are acceptable if done within 14 days before first study treatment dose).
* Severe illness or organ dysfunction involving the kidney, liver or other organ system (e.g. active uncontrolled infection , unstable angina pectoris or history of severe congestive heart failure, clinically unstable cardiac disease or pulmonary disease), which in the opinion of the investigator would interfere with the evaluation of the safety of the study treatment
* Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-11-06 (Actual); Primary Completion 2016-12-16 (Actual); Study Completion 2016-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (14):
- France (2):
  - 1230.33.33002 Boehringer Ingelheim Investigational Site, Marseille
  - 1230.33.33001 Boehringer Ingelheim Investigational Site, Paris
- Germany (12):
  - 1230.33.49011 Boehringer Ingelheim Investigational Site, Berlin
  - 1230.33.49002 Boehringer Ingelheim Investigational Site, Dresden
  - 1230.33.49001 Boehringer Ingelheim Investigational Site, Düsseldorf
  - 1230.33.49005 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 1230.33.49004 Boehringer Ingelheim Investigational Site, Freiburg im Breisgau
  - 1230.33.49010 Boehringer Ingelheim Investigational Site, Hamburg
  - 1230.33.49008 Boehringer Ingelheim Investigational Site, Hanover
  - 1230.33.49012 Boehringer Ingelheim Investigational Site, Kassel
  - 1230.33.49014 Boehringer Ingelheim Investigational Site, Leipzig
  - 1230.33.49009 Boehringer Ingelheim Investigational Site, Mannheim
  - 1230.33.49006 Boehringer Ingelheim Investigational Site, München
  - 1230.33.49003 Boehringer Ingelheim Investigational Site, Ulm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial had 2 parts.
Pre-assignment Details: Part 1:Starting dose of volasertib 250 mg administered on Day1 and Day15.The dose was escalated in 50 mg steps up to 300 mg.Flat dosing in Part 1. Part 2:volasertib dosing on Day1 in schedule A, on Day7 in schedule B, on Day1+ Day7 in schedule C.Body surface area (BSA) adapted dosing in Part 2. In each cycle, azacitidine was given from Day1 to 7
Groups:
- Volasertib 250 mg + Azacitidine (Escalation Cohort)-Part 1: Patients were intravenously administered escalating dose of volasertib 250 milligram (mg) (Volasertib (BI 6727), solution for infusion) on Day 1+15 (28-day cycle) combined with subcutaneous administration of Azacitidine (powder for reconstitution of an injection suspension) 75 milligram / square meter (mg/m2) once daily on Days 1 to 7 (28- day cycle)
- Volasertib 300 mg + Azacitidine (Escalation Cohort)- Part 1: Patients were intravenously administered escalating dose of volasertib 300 mg (Volasertib (BI 6727), solution for infusion) on Day 1+15 (28-day cycle) combined with subcutaneous administration of Azacitidine (powder for reconstitution of an injection suspension) 75 mg/m2 once daily on Days 1 to 7 (28-day cycle)
- Volasertib 250 mg + Azacitidine (Expansion Cohort)- Part 1: Patients were intravenously administered volasertib 250 mg (Volasertib (BI 6727), solution for infusion) on Day 1+15 (28-day cycle) combined with subcutaneous administration of Azacitidine (powder for reconstitution of an injection suspension) 75 mg/m2 once daily on Days 1 to 7 (28-day cycle) in the expansion cohort
- Volasertib 170 mg/m2 + Azacitidine (Escalation Cohort)- Part 2: Patients were intravenously administered escalating dose of volasertib 170 mg/m2 (Volasertib (BI 6727), solution for infusion) on Day 7 combined with subcutaneous administration of Azacitidine (powder for reconstitution of an injection suspension) 75 mg/m2 once daily on Days 1 to 7 (28-day cycle)
- Volasertib 110 mg/m2 + Azacitidine (Escalation Cohort)- Part 2: Patients were intravenously administered escalating dose of volasertib 110 mg/m2 (Volasertib (BI 6727), solution for infusion) on Day1 and Day 7 combined with subcutaneous administration of Azacitidine (powder for reconstitution of an injection suspension) 75 mg/m2 once daily on Days 1 to 7 (28-day cycle)
Period: Overall Study
Arm/Group | Volasertib 250 mg + Azacitidine (Escalation Cohort)-Part 1 | Volasertib 300 mg + Azacitidine (Escalation Cohort)- Part 1 | Volasertib 250 mg + Azacitidine (Expansion Cohort)- Part 1 | Volasertib 170 mg/m2 + Azacitidine (Escalation Cohort)- Part 2 | Volasertib 110 mg/m2 + Azacitidine (Escalation Cohort)- Part 2
Started | 6 | 6 | 1 | 2 | 1
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 6 | 1 | 2 | 1
Not completed — Adverse Event | 4 | 2 | 0 | 0 | 1
Not completed — Progressive disease / relapse | 0 | 1 | 0 | 1 | 0
Not completed — Other reason | 1 | 2 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): All entered patients receiving ≥1 dose of study medication were included in the TS
Groups:
- Total: Total of all reporting groups
Arm/Group | Volasertib 250 mg + Azacitidine (Escalation Cohort)-Part 1 | Volasertib 300 mg + Azacitidine (Escalation Cohort)- Part 1 | Volasertib 250 mg + Azacitidine (Expansion Cohort)- Part 1 | Volasertib 170 mg/m2 + Azacitidine (Escalation Cohort)- Part 2 | Volasertib 110 mg/m2 + Azacitidine (Escalation Cohort)- Part 2 | Total
Number analyzed (Participants) | 6 | 6 | 1 | 2 | 1 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.5 (8.2) | 69.2 (7.7) | 60.0 (NA) — One patient in this group | 64.5 (13.4) | 81.0 (NA) — One patient in this group | 68.9 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 0 | 1 | 3
  Male | 5 | 5 | 1 | 2 | 0 | 13

OUTCOME MEASURES:

1. Primary Outcome: Determination of the Maximum Tolerated Dose (MTD) Based on the Occurrence of Dose-limiting Toxicity (DLT) in Cycle 1
Description: The primary objective of the dose-escalation part of this study was to determine the MTD of volasertib in combination with azacitidine. The MTD was to be identified based on the DLT information collected during the first treatment cycle of each dosing schedule. DLT was defined as a non-haematological drug-related toxicity of Common Terminology Criteria for Adverse Events (CTCAE) grade ≥3. The MTD corresponded to the highest dose of volasertib and azacitidine at which the incidence of DLT was ≤17% (i.e. 1/6 patients) during Cycle 1.
  The planned dose escalation schedules of Part 2 were not completed because the trial was prematurely discontinued. Hence, a final conclusion of the MTD of volasertib in combination with azacitidine cannot be drawn in this trial.
  Number of patients with DLT in cycle 1 in escalation part is presented to determine MTD.
Time Frame: 4 weeks
Population: MTD set: The MTD set was used for the first treatment cycle (Cycle 1) analysis and excluded any treated patients that missed any dose of trial medication in Cycle 1 for reasons other than DLT
Measure: Number; unit: Milligram (mg)
Arm/Group | Volasertib 250 mg + Azacitidine (Escalation Cohort)-Part 1 | Volasertib 300 mg + Azacitidine (Escalation Cohort)- Part 1 | Volasertib 170 mg/m2 + Azacitidine (Escalation Cohort)- Part 2 | Volasertib 110 mg/m2 + Azacitidine (Escalation Cohort)- Part 2
Number analyzed (Participants) | 6 | 5 | 1 | 1
Milligram (mg) | NA — Final conclusion of the MTD of volasertib in combination with azacitidine could not be drawn in this trial. | NA — Final conclusion of the MTD of volasertib in combination with azacitidine could not be drawn in this trial. | NA — Final conclusion of the MTD of volasertib in combination with azacitidine could not be drawn in this trial. | NA — Final conclusion of the MTD of volasertib in combination with azacitidine could not be drawn in this trial.

2. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLT) in Cycle 1
Description: Number of participants with Dose Limiting Toxicities (DLT) in Cycle 1 (escalation part to determine MTD) is presented .
Time Frame: 4 weeks
Population: MTD set
Measure: Number; unit: participants
Arm/Group | Volasertib 250 mg + Azacitidine (Escalation Cohort)-Part 1 | Volasertib 300 mg + Azacitidine (Escalation Cohort)- Part 1 | Volasertib 170 mg/m2 + Azacitidine (Escalation Cohort)- Part 2 | Volasertib 110 mg/m2 + Azacitidine (Escalation Cohort)- Part 2
Number analyzed (Participants) | 6 | 5 | 1 | 1
participants | 1 | 1 | 0 | 1

3. Secondary Outcome: Percentage of Patients With Objective Response (OR)
Description: OR was defined as best overall response of complete remission (CR) or partial remission (PR) defined according to the International Working Group (IWG) 2006 criteria.
  Complete remission (CR):
  * Bone marrow: <5 % myeloblasts with normal maturation of all cell lines*
  * Persistent dysplasia will be noted*
  * Peripheral blood:
  * hemoglobin (Hgb) > 11 Grams Per Decilitre (g/dL)
  * Platelets >100 x 109/L
  * Neutrophils > 1.0 x 109/L
  * Blasts 0 % *Dysplastic changes should consider the normal range of dysplastic changes
  Partial remission (PR):
  All CR criteria if abnormal before treatment except:
  * Bone marrow blasts decreased by >50% to pre-treatment but still >5%
  * Cellularity and morphology not relevant
Time Frame: From randomisation until data cut-off (16Dec2016); up to 159 weeks
Population: Efficacy set (ES): All the treated patients without any protocol violations related to efficacy
Measure: Number; unit: percentage of participants
Arm/Group | Volasertib 250 mg + Azacitidine (Escalation Cohort)-Part 1 | Volasertib 300 mg + Azacitidine (Escalation Cohort)- Part 1 | Volasertib 250 mg + Azacitidine (Expansion Cohort)- Part 1 | Volasertib 170 mg/m2 + Azacitidine (Escalation Cohort)- Part 2 | Volasertib 110 mg/m2 + Azacitidine (Escalation Cohort)- Part 2
Number analyzed (Participants) | 6 | 5 | 1 | 2 | 1
percentage of participants | 33.3 | 20.0 | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: From randomisation until data cut-off (16Dec2016); up to 159 weeks
Arm/Group | Volasertib 250 mg + Azacitidine (Escalation Cohort)-Part 1 | Volasertib 300 mg + Azacitidine (Escalation Cohort)- Part 1 | Volasertib 250 mg + Azacitidine (Expansion Cohort)- Part 1 | Volasertib 170 mg/m2 + Azacitidine (Escalation Cohort)- Part 2 | Volasertib 110 mg/m2 + Azacitidine (Escalation Cohort)- Part 2
Serious Adverse Events (participants affected / at risk) | 6/6 | 2/6 | 0/1 | 0/2 | 1/1
Other Adverse Events (participants affected / at risk) | 6/6 | 5/6 | 1/1 | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Volasertib 250 mg + Azacitidine (Escalation Cohort)-Part 1 (N=6) | Volasertib 300 mg + Azacitidine (Escalation Cohort)- Part 1 (N=6) | Volasertib 250 mg + Azacitidine (Expansion Cohort)- Part 1 (N=1) | Volasertib 170 mg/m2 + Azacitidine (Escalation Cohort)- Part 2 (N=2) | Volasertib 110 mg/m2 + Azacitidine (Escalation Cohort)- Part 2 (N=1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Volasertib 250 mg + Azacitidine (Escalation Cohort)-Part 1 (N=6) | Volasertib 300 mg + Azacitidine (Escalation Cohort)- Part 1 (N=6) | Volasertib 250 mg + Azacitidine (Expansion Cohort)- Part 1 (N=1) | Volasertib 170 mg/m2 + Azacitidine (Escalation Cohort)- Part 2 (N=2) | Volasertib 110 mg/m2 + Azacitidine (Escalation Cohort)- Part 2 (N=1)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 1 | 0
Cyclic neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 3 | 1 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 5 | 1 | 1 | 1
Cardiac valve disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Thyroid mass (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0
Scleral haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 2 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 1 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 2 | 0 | 2 | 0
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 1 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 1 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 2 | 0 | 0 | 0
Feeling cold (General disorders) | 0 | 0 | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1 | 1
Inflammation (General disorders) | 1 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 1 | 0 | 0 | 1 | 0
Oedema (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 1 | 0 | 0 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 1 | 0 | 0
Hepatic lesion (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Haematoma infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infected bite (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Tooth avulsion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Blood creatine increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 1 | 1 | 1 | 1
Blood folate decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Body temperature increased (Investigations) | 0 | 0 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 1 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Growing pains (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0
Libido disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Renal disorder (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0 | 0
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 1 | 1 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The sponsor discontinued the development of volasertib on 25 Nov 2016 and this trial was discontinued on 16 Dec 2016 for non-clinical reasons. The number of patients enrolled in Part 2 of the study was too small for a meaningful analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.